CLINICAL TRIAL: NCT00321451
Title: Behavioral Insomnia Therapy With Fibromyalgia
Brief Title: Cognitive Behavioral Insomnia Therapy for Individuals With Fibromyalgia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00011861; R01AR052368 (NIH)
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Fibromyalgia; Sleep Initiation and Maintenance Disorders
Keywords: insomnia; cognitive behavior therapy
MeSH Terms: conditions — Fibromyalgia; Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia
- 2 (Sham Comparator)
  Interventions: Behavioral: Pseudo-desensitization procedure
- 3 (Active Comparator)
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia — 4 biweekly outpatient sessions with sleep psychologist
  Arms: 1
Behavioral: Pseudo-desensitization procedure — 4 biweekly outpatient visits with sleep psychologist
  Arms: 2
Other: Usual care — 3 outpatient visits with study physician
  Arms: 3

SUMMARY:
Fibromyalgia (FM) is a common and chronic disorder characterized by widespread muscle pain, fatigue, and multiple tender points. The majority of individuals with FM report sleep problems, including delayed sleep onset, extended awakenings, and non-restorative sleep. These sleep disturbances may worsen FM-related pain, fatigue, low mood, and low energy. The purpose of this study is to evaluate the effectiveness of cognitive behavioral insomnia therapy in reducing sleep disturbances and improving other FM-related symptoms.

DETAILED DESCRIPTION:
FM is a debilitating condition that can lead to impaired occupational and social functioning, disability, and increased health care utilization. FM symptoms vary among individuals, but they typically include chronic widespread pain, persistent daytime fatigue, sleep disturbances, low mood, and loss of stamina. The cause of FM remains unknown, and current treatment involves symptom-focused interventions such as antidepressants, behavioral stress management, coping skills training, and exercise programs. However, there are no interventions specifically designed to reduce sleep disturbances in people with FM.

Past research has shown that individuals with FM experience the same behavioral and psychological factors that individuals suffering from insomnia experience. Cognitive behavioral insomnia therapy, a form of psychotherapy that aims to eliminate factors that disrupt sleep, may prove useful for people with FM. The purpose of this study is to evaluate the effectiveness of cognitive behavioral insomnia therapy in reducing sleep disturbances and improving FM-related pain, fatigue, mood, and quality of life among individuals with FM. The study will also examine the use of sleep electroencephalogram (EEG) as a means to measure improvements in FM symptoms.

This study will last about 9 months and will include approximately 16 study visits. An initial 2-week screening period will include a physical examination, blood collection, a mental status exam, a tender-point exam, a sleep history questionnaire, and structured sleep and psychiatric interviews. Participants will complete a 1-week sleep log and one overnight polysomnogram test, in which several body functions (e.g., brain activity, eye movement, heart rate, etc.) are recorded. If an FM diagnosis is confirmed, an additional 2-week assessment period will take place, followed by an 8-week treatment period. During treatment, participants will be randomly assigned to one of the following three treatment groups: 1) usual FM care (medical advice and medication prescription), 2) usual FM care plus psychological treatment to decrease insomnia, and 3) usual FM care plus placebo psychological treatment to decrease insomnia. Groups 2 and 3 will attend four bi-weekly individual therapy sessions with a sleep psychologist. Participants will meet with a rheumatologist at least once. Throughout treatment, nightly sleep logs and medication questionnaires will be completed, and participants will wear a wrist-watch sized device that will record their day- and night-time activity. A therapy evaluation questionnaire will be completed during the first and last weeks of treatment and an outcome questionnaire packet will be completed after 4 weeks of treatment. All participants will be evaluated following the end of treatment and again 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Reside in or around Durham, NC
* History of insomnia complaints for more than 1 month
* Diagnosis of primary FM
* Diagnosis of insomnia

Exclusion Criteria:

* Terminal illness or acute serious medical illness
* Secondary FM or condition other than FM that seriously compromises sleep
* Current psychiatric illness or currently suicidal
* Substance abuse or dependence
* Other primary sleep disorder (e.g., sleep apnea or restless legs syndrome)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2006-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Total wake time | Measured immediately and 6 months post-treatment
Total sleep time | Measured immediately and 6 months post-treatment
Sleep efficiency | Measured immediately and 6 months post-treatment

SECONDARY OUTCOMES:
Sleep onset latency | Measured immediately and 6 months post-treatment
Wake time after sleep onset | Measured immediately and 6 months post-treatment
Score on an insomnia rating scale | Measured immediately and 6 months post-treatment
Score on a fatigue rating scale | Measured immediately and 6 months post-treatment
Score on a mood rating scale | Measured immediately and 6 months post-treatment
Subjective pain ratings | Measured immediately and 6 months post-treatment
Score on a health-related quality of life scale | Measured immediately and 6 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jack D. Edinger, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Edinger JD, Wohlgemuth WK, Krystal AD, Rice JR. Behavioral insomnia therapy for fibromyalgia patients: a randomized clinical trial. Arch Intern Med. 2005 Nov 28;165(21):2527-35. doi: 10.1001/archinte.165.21.2527. PMID 16314551